CLINICAL TRIAL: NCT02806622
Title: Comparison of Hip Range of Motion Values Among NCAA Division II Collegiate Athletes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: California State University, Dominguez Hills (Other)
Responsible Party: Principal Investigator, Scott Cheatham, Assistant Professor, California State University, Dominguez Hills
Other Study IDs: 16-208
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Disorder of Hip Joint
Keywords: Sports; University; Lower Extremity; Hip Joint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Division II Collegiate Athletes: Student athletes (18-45) currently enrolled and participating on a sports team.

SUMMARY:
The purpose of this study is to compare hip passive range of motion (ROM) among division II collegiate athletes in order to obtain normative data for future research. The investigators hypothesize that there will be a difference in passive hip ROM among the different genders and sports.

DETAILED DESCRIPTION:
Currently there is no normative data for hip passive ROM in apparently healthy NCAA division II collegiate athletes. This study will be the first study to develop preliminary normative data of hip passive ROM.

One hundred (N=100) student athletes (18-45 years) from California State University Dominguez Hills (CSUDH) will be recruited for this study via convenience sampling. Data collection will take place in the CSUDH sports medicine laboratory. Prior to testing, participants will fill out a screening questionnaire with questions that represent the exclusion criteria which will be used to determine ineligibility for this study.

Prior to participant recruitment and enrollment, a pilot study will be done on 10 participants to establish rater reliability using the methods mentioned below. After acceptable reliability is achieved, recruitment and enrollment will continue.

Participants who meet the inclusion criteria and consent to participate will be enrolled in the study. Participants will read and sign a CSUDH approved consent form prior to beginning data collection. Following consent, participants will also fill out a questionnaire to provide demographic information which includes age, height, weight, and leg dominance.

Following completion of the paperwork, all participants will undergo testing which will be conducted between the hours of 8am and 4pm. Each data collection session will last for approximately 20 minutes. Bilateral hip passive ROM data will be collected using the Noraxon computerized motion system. Participants will be lying in different positions on an examination table while the hip joints and lower extremities are moved into different positions and measured by the device which will touch the skin. Data will be collected and monitored by the examiner using the computerized system. The data collection protocol for both lower extremities are as follows:

1. Supine measures (passive): hip external rotation, hip internal rotation
2. Rest: 5-minute delay
3. Seated measures (passive): hip external rotation, hip internal rotation
4. Rest: 5-minute delay
5. Prone measurements (passive): hip external rotation, hip internal rotation

Collected data will be transferred to SPSS v.22 (IBM SPSS, Chicago, IL). Means,standard deviations, 95% confidence intervals (95% CI), and ranges for participant descriptive data will be calculated. Passive Hip ROM values will be presented using degrees and percentages. Athlete gender and sport differences will be calculated using the ANOVA statistic. The p-value will be considered significant at the .05 level using a two-tailed test (α2 =.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy student collegiate athletes

Exclusion Criteria:

* Presence of musculoskeletal, systemic or metabolic diseases that would affect lower extremity joint ROM or muscle function
* Presence of any current or past muscle or joint pathology of the hip, knee, and/or ankle that would affect lower extremity joint ROM or muscle function
* Inability to avoid exercise 4 hours prior to testing
* Inability to avoid medications that may affect the outcome of lower extremity joint ROM or muscle function

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Division II collegiate athletes (18-45) currently enrolled in school and participating on a sports team.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Hip Joint Internal and External Rotation ROM | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Cheatham, DPT, PhD, Principal Investigator — California State University, Dominguez Hills

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shimamura KK, Cheatham S, Chung W, Farwell D, De la Cruz F, Goetz J, Lindblom K, Powers D. Regional interdependence of the hip and lumbo-pelvic region in divison ii collegiate level baseball pitchers: a preliminary study. Int J Sports Phys Ther. 2015 Feb;10(1):1-12. PMID 25709857
- [Background] Prather H, Harris-Hayes M, Hunt DM, Steger-May K, Mathew V, Clohisy JC. Reliability and agreement of hip range of motion and provocative physical examination tests in asymptomatic volunteers. PM R. 2010 Oct;2(10):888-95. doi: 10.1016/j.pmrj.2010.05.005. PMID 20970757
- [Background] Krause DA, Hollman JH, Krych AJ, Kalisvaart MM, Levy BA. Reliability of hip internal rotation range of motion measurement using a digital inclinometer. Knee Surg Sports Traumatol Arthrosc. 2015 Sep;23(9):2562-7. doi: 10.1007/s00167-014-3096-0. Epub 2014 Jun 11. PMID 24912575
- [Background] Roach S, San Juan JG, Suprak DN, Lyda M. Concurrent validity of digital inclinometer and universal goniometer in assessing passive hip mobility in healthy subjects. Int J Sports Phys Ther. 2013 Oct;8(5):680-8. PMID 24175147